CLINICAL TRIAL: NCT03218774
Title: Does Participating in a Supervised Fitness Program Extend the Benefits of Episodic Physical Therapy More Than a Home Exercise Program for Adults With Cerebral Palsy?
Brief Title: Supervised Fitness Program for Adults With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Sheltering Arms Physical Rehabilitation Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HM20009344
Record Dates: First submitted 2017-07-12; First posted 2017-07-17 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to group assignment. It is not possible to blind the participants or the care providers.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Group (Other)
  Interventions: Behavioral: Home Exercise Group
- Center Group (Experimental)
  Interventions: Behavioral: Fitness Center Group

INTERVENTIONS:
Behavioral: Home Exercise Group — The Home group will meet with an exercise professional once and be given a home exercise program to complete 3 to 5 times per weeks at home.
  Arms: Home Group
Behavioral: Fitness Center Group — The Center group will be given an exercise program, a membership to a community fitness gym where they will be asked to exercise 3-5 times per week, and will be provided with 6 individual personal training sessions.
  Arms: Center Group

SUMMARY:
The purpose of this study is to compare the effectiveness of 2 community intervention approaches to maintain community mobility and walking speed in adults with cerebral palsy who have previously completed an 8 week course of physical therapy.

DETAILED DESCRIPTION:
The proposed study will address the lifelong need for fitness in adults with cerebral palsy compared to individuals provided with a home exercise program at the end of their individualized physical therapy, individuals in the fitness group will…

Primary Hypothesis:

1. Have higher Pediatric Evaluation of Disability Inventory Computer Adapted Test (PEDICAT) scores at the +12 weeks post intervention visit
2. Increase their PEDICAT scores across the study period, while the home fitness group will decrease performance on the PEDICAT.
3. Complete the Timed Up and Go (TUG) more quickly at +12 weeks post intervention

   Secondary Hypothesis (study not powered for these variables):
4. Walk further on the Six Minute Walk Test (6MWT) at the +12 weeks post intervention visit

ELIGIBILITY:
Inclusion Criteria:

* Adults with cerebral palsy Gross Motor Function Classification System (GMFCS) level I, II, or III
* Completion of episode of physical therapy provided by the Developmental Disabilities program at Sheltering Arms within the one month prior to the baseline assessment
* Lives within the community in their own home or group housing

Exclusion Criteria:

* GMFCS level IV or V
* Unable to follow two-step directions
* Adults who have a medical or legal power of attorney who sign their health authorization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Change in Pediatric Evaluation of Disability Inventory - Computer Adaptive Testing Version (PEDICAT) score | Baseline, 4 weeks, 8 weeks, 12 weeks
  The PEDI-CAT assesses function in 4 domains: Daily Activity, Mobility, Social/Cognitive, Responsibility
Change in Timed Up and Go (TUG) score | Baseline, 4 weeks, 8 weeks, 12 weeks
  Mobility assessment measuring amount of time it takes for participant to get up from chair, walk to a line on the floor at a normal pace, and return to a seated position

SECONDARY OUTCOMES:
Change in six-minute walk test (6MWT) | Baseline, 4 weeks, 8 weeks, 12 weeks
  measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface

CONTACTS AND LOCATIONS:
Overall Officials: Stacey C Dusing, Ph.D., PT, Principal Investigator — Virginia Commonwealth University
Locations (2):
- United States (2):
  - Sheltering Arms, Mechanicsville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia